CLINICAL TRIAL: NCT05899920
Title: Clinical One-stage Controlled Study of reSistant Arterial Hypertension for the desiGning of a personAlized Approach to Therapy
Acronym: SAGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SAGA-01
Record Dates: First submitted 2023-05-02; First posted 2023-06-12 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Resistant Arterial Hypertension
Keywords: antihypertensive drugs; concentration; HPLC MS/MS
MeSH Terms: interventions — Pharmacokinetics; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled arterial hypertension (Active Comparator): Controlled arterial hypertension according the results of 24-hour blood pressure monitoring.
  Blood samples will be taken for pharmacokinetics and pharmacogenetics
  Interventions: Diagnostic Test: Blood samples will be taken for pharmacokinetics and pharmacogenetics
- Uncontrolled arterial hypertension (Experimental): Uncontrolled arterial hypertension according the results of 24-hour blood pressure monitoring.
  Blood samples will be taken for pharmacokinetics and pharmacogenetics
  Interventions: Diagnostic Test: Blood samples will be taken for pharmacokinetics and pharmacogenetics

INTERVENTIONS:
Diagnostic Test: Blood samples will be taken for pharmacokinetics and pharmacogenetics — To assess antihypertensive drugs concentration (lisinopril, valsartan, amlodipine, indapamide

SUMMARY:
This study was planned to assess the concentration of antihypertensive drugs in the blood plasma in patients with controlled and uncontrolled arterial hypertension. Methods: it is planned to include patients with arterial hypertension taking 3 antihypertensive drugs (indapanide, lisinopril or valsartan, amlodipine). Based on the results of 24-hour blood pressure monitoring, the patients will be randomized into two groups: The first group - the patients with controlled AH; The second group - the patients with uncontrolled AH. Venous blood was taken in both groups of the patients in the morning before and 2 hours after taking drugs to assess the concentration of lisinopril, amlodipine, valsartan and indapamide. Concentation of assesed antihypertensive drugs will be compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* An established diagnosis of AH based on the Clinical Guidelines "Arterial hyperten-sion in adults", approved by the Scientific and Practical Council of the Ministry of Health of the Russian Federation, 2020;
* Mandatory patient compliance with recommendations for lifestyle modification in accordance with the Clinical Guidelines "Arterial hypertension in adults", approved by the Scientific and Practical Council of the Ministry of Health of the Russian Federation, 2020 .
* Regular administration of any two antihypertensive drugs (lisinopril, amlodipine, valsartan) in combination with indapamide for a month, possibly in fixed combinations, in stable dosages;
* Fertile female patients must use proper methods of contraception throughout the study period.

Exclusion Criteria:

* Patient's connection with the organization or conducting of the study;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-11-11 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of lisinopril, valsartan, amlodipin, indapamide, metoprolol | day 1
  Number of Participants with antihypertensive drug concentraion below the limit of quantitative determination

CONTACTS AND LOCATIONS:
Locations (1):
- Ryzan State Medical University, Ryazan, Russia